CLINICAL TRIAL: NCT04728568
Title: Exploratory Study of PD-1 Neoadjuvant Treatment of Recurrent Meningioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 320.6750.2020-10-02
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Meningioma, Malignant
Keywords: Sintilimab
MeSH Terms: conditions — Meningioma | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab (Experimental): Sintilimab will be administered every 3 weeks Sintilimab will be administered through IV infusion
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab binds to PD-1, an inhibitory signaling receptor expressed on the surface of activated T cells, and blocks the binding to and activation of PD-1 by its ligands, which results in the activation of T-cell-mediated immune responses against tumor cells
  Other Names: Sintilimab Injection

SUMMARY:
This research study is studying a drug as a possible treatment for High Grade Meningioma.

DETAILED DESCRIPTION:
Meningioma is one of the most common primary intracranial tumors, accounting for 13% to 26% of all intracranial tumors. Although most meningiomas are benign tumors and can be cured by surgical resection, more than 20% of WHO II (atypical) and about 3% of WHO III meningiomas are more likely to have local recurrence after initial treatment , And the lifetime is poor. The immunotherapy represented by PD-1 has achieved remarkable efficacy in the treatment of solid tumors, but the application of PD-1 in recurrent meningioma is rarely reported. The study found that the expression of PD-L1 mRNA and protein in high-grade meningioma cells increased, and the total number of T cells, including CD4+ and CD8+ cells, was significantly reduced, suggesting an inhibitory tumor immune microenvironment. Recent studies have shown that giving patients anti-PD-1 antibody immunotherapy prior to conventional treatment can improve the pathological response, enable the body to produce an enhanced and sustained anti-tumor immune response, and form a tumor microenvironment conducive to immunotherapy. Therefore, giving PD-1 antibody before surgery is a new idea for the treatment of meningiomas. This project aims to investigate whether patients with recurrent meningioma will change their immune function and prolong survival after preoperative PD-1 antibody treatment. It is planned to use flow cytometry, multiple immunofluorescence histochemistry technology, T cell receptor sequencing, etc to detect the changes in the patient's immune function before and after treatment, observe the pathological remission rate of PD-1 monoclonal antibody neoadjuvant treatment of recurrent meningioma, and identify potential response biomarkers, and conduct in-depth discussions on this treatment plan to further determine the treatment mode Clinical value and specific mechanism of action in order to improve the clinical treatment level of patients with recurrent meningioma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as a patient with WHO grade III recurrent meningioma
* Age ≥ 18 years
* Kps≥70
* able to accept second surgery
* ECOG Performance Status < 2
* Glucocorticoid dosage dexamethasone ≤5mg/ day or equivalent dose

Exclusion Criteria:

* Participants who have had chemotherapy, targeted small molecule therapy or study therapy within 14 days of protocol treatment, or those who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants who have a diagnosis of an immunodeficiency.
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone >2mg/day or bioequivalent within 7 days of initiating therapy.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent. Unable to undergo brain MRI.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Every 6 weeks, up to 6 months
  Contrast-enhanced cranial MRI will be performed every 6 weeks. PFS6 is defined as not having progressive disease or death within six months of the first day of treatment. Contrast-enhanced cranial magnetic resonance imaging (MRI) will be performed every 6 weeks.

SECONDARY OUTCOMES:
Overall Survival | 6 months and 12 months
  The distributions of overall survival will be summarized using the method of Kaplan-Meier. The follow-up of patients who are alive at the time of analysis will be censored at the date of last assessment of vital status. Median OS will be presented and accompanied by 90% confidence intervals estimated using log(-log(survival)) methodology. Survival point estimates at 3 and 6 months will also be presented with confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Chen, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing TianTan Hospital, Beijing, Beijing Municipality, China